CLINICAL TRIAL: NCT01728285
Title: A Multicentric Open Randomised, Cross-over Phase III Trial Assessing the Treatment Compliance With GRAZAX® in Subjects With Seasonal Grass Pollen Induced Rhinoconjunctivitis
Brief Title: Compliance to the Treatment With GRAZAX® Tablets in Patients With Seasonal Grass Pollen Rhinoconjunctivitis
Acronym: GT-17
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GT-17 ITALY; 2006-004820-35 (EudraCT Number)
Record Dates: First submitted 2012-11-02; First posted 2012-11-19 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Allergic Rhinitis; Grass Allergy
Keywords: specific allergen immunotherapy; sublingual immunotherapy; allergen tablets; compliance; electronic compliance device
MeSH Terms: conditions — Rhinitis, Allergic; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electronic compliance device (Active Comparator): Patients with grass allergy treated with allergen specific immunotherapy (GRAZAX®) using an electronic compliance device (Memozax®)
  Interventions: Device: Electronic compliance device (Memozax®)
- No electronic compliance device (No Intervention): Patients with grass allergy treated with allergen specific immunotherapy (GRAZAX®) without any electronic compliance device (Memozax®)

INTERVENTIONS:
Device: Electronic compliance device (Memozax®) — An electronic compliance device is distributed to patients allocated to the active arm
  Arms: Electronic compliance device

SUMMARY:
Adherence to treatment is crucial to the efficacy of sublingual immunotherapy of allergic diseases. GRAZAX® is a registered drug in Europe, with established efficacy in the treatment of allergic rhinitis, which has to be taken daily by patients. This study was aimed to establish if a device with the characteristics of a mechanical dispenser (Memozax®) could improve adherence to treatment in subjects with hay fever due to allergy to grass

ELIGIBILITY:
Inclusion Criteria:

* A clinical history of grass pollen-induced allergic rhinoconjunctivitis (with or without asthma) having received treatment during the previous grass pollen season.
* Positive skin prick test (SPT) response (wheal diameter ≥3mm) to Phleum pratense
* Positive specific IgE against Phleum pratense (IgE titer > class 2)

Exclusion Criteria:

* Clinical history of chronic sinusitis during the last 2 years or of symptomatic perennial or seasonal allergic rhinitis and/or asthma having received regular medication, due to another allergen during - or potentially overlapping - the grass pollen season.
* Clinical history of severe asthma (GINA Step 4 and children with Forced Expiratory Volume in 1 second (FEV1) < 80% of expected value after treatment with inhaled corticosteroids and short-acting β2 agonists)
* Previous treatment by immunotherapy with grass pollen allergen or any other allergen within the previous 5 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2007-03; Primary Completion 2009-06 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To evaluate if compliance with grass Allergy Immunotherapy Tablet can be increased by providing an electronic compliance device (CED) (Memozax; a tablet-container with a programmable daily acoustic alarm) | up to 1 year per patient
  To evaluate if compliance of once daily dosing with Grazax in adult subjects with grass pollen induced allergic rhinoconjunctivitis can be increased by providing patients with an electronic compliance device. Compliance in the two groups (with Memozax and without Memozax) was evaluated by tablet counts

SECONDARY OUTCOMES:
Impact of GRAZAX® treatment on QoL as compared to previous season | up to 1 year per patient
  To evaluate after one-year treatment with Grazax tablets the impact on quality of life in comparison with previous pollen seasons
Impact of GRAZAX® treatment on allergy symptoms as compared to previous season | up to 1 year per patient
  To evaluate after one-year treatment with Grazax tablets the impact on symptom score in comparison with previous pollen seasons
Impact of GRAZAX® on treatment acceptance as compared to previous season | up to 1 year per patient
  To evaluate after one-year treatment with Grazax tablets the impact on patient's acceptance in comparison with previous pollen seasons
Recording of all adverse events and serious adverse events | up to 1 year per patient
  The safety assessments included recording of all adverse events (AE) and serious adverse events (SAE) findings from physical examinations and from vital signs

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, PV, Italy

REFERENCES:
- [Result] Alesina R, Milani M, Pecora S. A multicenter, randomized, parallel-group trial assessing compliance, tolerability, safety, and efficacy to treatment with grass allergy tablets in 261 patients with grass pollen rhinoconjunctivitis. J Allergy (Cairo). 2012;2012:673502. doi: 10.1155/2012/673502. Epub 2011 Nov 9. PMID 22131999